CLINICAL TRIAL: NCT02600637
Title: Evaluation of Wellness Programs for Brain-Injured Individuals
Brief Title: Wellness Programs for Brain-Injured Individuals
Acronym: WPBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1893-P
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Depression; Anxiety; Stroke
Keywords: stroke; depression; anxiety; mindfulness; meditation
MeSH Terms: conditions — Depression; Anxiety Disorders; Stroke | interventions — Meditation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBSR (Experimental): Mindfulness-based Stress Reduction program
  Interventions: Behavioral: MBSR
- Education (Active Comparator): Educational group program
  Interventions: Behavioral: Brain Health class

INTERVENTIONS:
Behavioral: MBSR — Mindfulness-based Stress Reduction is an 8-week course designed to teach a number of mindfulness techniques to help improve stress- and depression-related symptoms.
  Other Names: Meditation
  Arms: MBSR
Behavioral: Brain Health class — An 8-week course on brain health will be administered to participants as an active control group.
  Other Names: Psychoeducation
  Arms: Education

SUMMARY:
Summary: Thousands of Veterans suffer a stroke every year, and these individuals often suffer emotional and cognitive changes that negatively affect their quality of life as well as their ability to recover. In addition to traditional rehabilitation such as physical and occupational therapy, a number of alternative treatments are now being studied for their ability to enhance patients' recovery following stroke. One of these treatments, Mindfulness-Based Stress Reduction or MBSR, involves an 8-week course that teaches individuals strategies such as breathing techniques, meditation, and movement therapy. The current pilot study proposes to teach MBSR to a group of Veterans with a history of stroke to determine whether this type of intervention is feasible, acceptable to patients, and shows preliminary evidence of beneficial effects on psychological and cognitive functioning. The investigators hope to find that MBSR is a useful, additional intervention that can improve Veterans' well-being and quality of life as they recover from stroke.

DETAILED DESCRIPTION:
Description: Stroke affects approximately 800,000 Americans every year, including thousands of Veterans, and is a leading cause of disability in the US. While many stroke patients receive rehabilitation during the acute and post-acute phases of stroke, many individuals suffer chronic deficits and have few options for continued treatment. A number of low-cost, alternative treatments are now being tested for their usefulness in treating neuropsychological deficits in chronic stroke patients. One of the best studied of these treatments is Mindfulness-Based Stress Reduction (MBSR), which involves an 8-week course led by a trained instructor. MBSR teaches individuals strategies for coping with their injury, such as meditation, breathing techniques, and sensory awareness. A handful of preliminary studies have shown that MBSR is effective in reducing symptoms of depression and anxiety in stroke patients, as well as enhancing performance on cognitive tasks. However, only a single randomized controlled trial of MBSR in stroke has been published to date, and that study suffered from a number of weaknesses such as the lack of an active control group. Moreover, no previous study has assessed the usefulness of MBSR for stroke in a Veteran population. Therefore, the current study proposes to undertake a rigorous, randomized controlled pilot study of MBSR in Veterans with a history of stroke, using an active control group, blinded examiners, and a 3-month follow-up session to determine whether any benefits of MBSR are long-lasting. For the study, 60 Veterans with a history of chronic stroke will be recruited: 30 patients will be randomly assigned to the MBSR intervention, and 30 patients will be assigned to a Brain Health education program, which will be matched to the MBSR group with respect to the instructor, number of hours of instruction, homework activities, and class size. A blinded examiner will complete a neuropsychological assessment of patients' emotional and cognitive status at three time points: 1) prior to the intervention, 2) following the intervention (within 1 week), and 3) three months later. The investigators will evaluate a number of feasibility factors in this pilot study, including patient recruitment and retention procedures, effectiveness of randomization and blinding measures, and patient acceptability. Preliminary evaluation of the MBSR intervention will test for clinically reliable improvements in anxiety and depressive symptomatology following the intervention, relative to the Brain Health group, as well as improvements on a cognitive test battery. It is also predicted that changes associated with the MBSR intervention will still be present at the 3-month follow-up assessment as well. The final objective of the current proposal is an exploratory aim to determine whether the site of a patient's stroke plays a role in their ability to benefit from MBSR. Previous research has suggested that left prefrontal cortex plays a critical role underlying the effects of MBSR. Thus, patients with and without left prefrontal involvement will be compared, and it is predicted that involvement of this brain region will modulate the observed effects. Such information could be used to target those Veterans who can most benefit from the proposed intervention. If successful, the investigators plan to execute a larger efficacy study to evaluate the magnitude of treatment effects associated with MBSR. Alternative interventions such as MBSR can provide low-cost, non-invasive rehabilitative treatments for chronic stroke that can improve Veterans' functional recovery and general sense of well-being.

ELIGIBILITY:
Inclusion Criteria:

* A history of a single, chronic right or left hemisphere stroke (> 6 months post-onset so that residual symptoms have stabilized)
* Age 20-80
* Native English proficiency
* At least mild level of depression and/or mild anxiety
* Language within normal limits so that language deficits will not interfere with the intervention

Exclusion Criteria:

* A pre-morbid neurologic history or history of schizophrenia spectrum and other psychotic disorders
* Bipolar disorders
* Depressive disorders with psychotic features (to avoid potential confounds in neuropsychological testing)
* Mini-Mental State Examination score <19 (suggesting moderate to severe cognitive impairment that is a contraindication in effectively participating in the MBSR intervention52)
* Recent substance abuse/dependence disorder (< 1 year)
* Acutely suicidal (defined below)
* Concurrent involvement in another rehabilitation program
* Significant visual or hearing disabilities that would preclude participating in the program
* Medical history, including pre-morbid neurologic and psychiatric history, will be assessed with a standard medical questionnaire during the initial interview session as well as a review of patients' VA medical records
* Medications will not be an exclusionary factor for participation but will be recorded and tracked via VA computerized medical record systems

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana V. Baldo, PhD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MBSR | Education
Started | 19 | 18
Completed | 14 | 13
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBSR | Education | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (12.0) | 67.3 (9.5) | 66 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 15 | 15 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 13 | 15 | 28
  black | 4 | 2 | 6
  asian | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Depression Score Change on Geriatric Depression Scale
Description: Determine whether the MBSR treatment has any effect on depression by comparing change scores (post-intervention minus pre-intervention) on the Geriatric Depression Scale (GDS) for MBSR versus Education control group. A negative change score indicates improvement in depressive symptomatology. Full score range possible on the GDS is 0-30, where 0 means no depression and 30 means severe depression.
Time Frame: Over the 8 week assessment period for each participant, up to a total of 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR | Education
Number analyzed (Participants) | 19 | 18
units on a scale | -.29 (3.2) | -1.46 (2.5)

2. Primary Outcome: Anxiety Score Change on State-Trait Anxiety Inventory Questionnaire
Description: Determine whether the MBSR treatment has any effect on anxiety by comparing change score (post-intervention minus pre-intervention) on State-Trait Anxiety Inventory (STAI) for MBSR versus Education control group. A negative change score indicates improvement in anxiety symptoms. Full range of scores on the STAI is 20-80, where 20 is minimal/no anxiety and 80 is severe anxiety.
Time Frame: Over the 8 week assessment period for each participant, up to a total of 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR | Education
Number analyzed (Participants) | 19 | 18
units on a scale | .57 (.21) | -2.31 (.7)

3. Secondary Outcome: Repeatable Battery for Assessment of Neuropsychological Status Battery Overall Cognitive Change Score
Description: Determine whether the MBSR treatment has any effect on overall cognitive performance by comparing the change score (post-intervention minus pre-intervention) in overall Cognitive standard score on RBANS for MBSR versus Education control group. Positive change score indicates improvement in overall cognitive performance. The possible range of standard scores on the RBANS is 40-154, where 40 is severely impaired cognition and 154 is superior range cognition.
Time Frame: Over the 8 week assessment period for each participant, up to a total of 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR | Education
Number analyzed (Participants) | 19 | 18
units on a scale | 7.69 (1.2) | 3.08 (.4)

ADVERSE EVENTS:
Time Frame: Over the 8 week assessment period for each participant, up to a total of 5 months
Description: did not differ
Arm/Group | MBSR | Education
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT02600637/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT02600637/SAP_001.pdf